CLINICAL TRIAL: NCT05547633
Title: Detection and Management of Sinusitis in a Single-center Prospective Cohort of Patients With Exudative AMD (SINE)
Acronym: SINE
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: RLX-2022-4
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: AMD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: sinusitis screening consultation — Questioning to look for suspicious anamnestic elements such as rhinorrhea, nasal obstruction, smell disorders, facial pain and clinical examination including nasofibroscopy.
  Patients with signs of sinusitis will be managed according to current recommendations (diagnostic imaging tests, medical treatment or even surgery if necessary).

SUMMARY:
An inflammatory component associated with AMD has been highlighted by genetic associations of predisposition to AMD, as well as by the recently demonstrated link between AMD and periodontitis.

Some patients followed at the Fondation Adolphe de Rothschild Hospital for wet AMD seemed to show an improvement of neovascular activity (less need for intravitreal injections of anti-VEGF) after treatment of their sinusitis.

The investigators would therefore like to assess the link between AMD and sinusitis, an infection close to the site of AMD.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient followed and treated for at least 2 years for bilateral neovascular form of age-related macular degeneration (AMD)
* At least one eye treated with ≥ 6 intravitreal injections during the year preceding preinclusion
* Express consent to participate in the study
* Affiliated with or beneficiary of a social security plan

Exclusion Criteria:

* Persons referred to in articles L1121-5 to L1121-8 of the CSP (corresponding to all protected persons: pregnant women, parturients, nursing mothers, persons deprived of liberty by judicial or administrative decision, minors, and persons under legal protection: guardianship or curatorship).
* Severe myopia (> 6 diopters)
* Patient already being treated for acute or chronic sinusitis
* History of central serous chorioretinopathy or diffuse retinal epitheliopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed at The Rothschild Hospital Foundation hospital for neovascular AMD receiving at least 6 intravitreal injections/year in at least one eye over the past 2 years.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Estimate the prevalence of sinusitis in patients with bilateral multi-injected neovascular AMD (≥ 6 intravitreal injections per year in at least one eye) | Day 0
  Percentage of patients with bilateral multiinjected neovascular AMD (≥6 intravitreal injections/year in at least one eye) with sinusitis following ENT consultation screening.
  Sinusitis is defined by nasofibroscopic abnormalities showing sinus pathology (inflammation, polyp, rhinorrhea) and/or scannographically confirmed sinus filling (some sinusitis is blocked and therefore not externalized).

SECONDARY OUTCOMES:
To compare, between patients screened and managed for sinusitis and those not requiring treatment for sinusitis, the evolution of the number of intravitreal injections | Month 15
  Comparison of the change in the number of intravitreal injections performed over a 1-year period before sinusitis screening and then over a 1-year period after completion of sinusitis treatment (for patients treated for sinusitis) or a 1-year period after the screening visit for patients not treated for sinusitis.
  If only one of the two eyes received 6 or more injections in the year before inclusion, the evolution of the number of injections for this eye will be considered. If both eyes received 6 or more injections in the year before inclusion, the eye with the most injections will be considered, if both eyes received the same number of injections the right eye will be considered by default.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Fondation A. de Rothschild, Paris, France